CLINICAL TRIAL: NCT06767150
Title: StrAtegies For Zoledronic Acid Post-dEnosumab Discontinuation in Postmenopausal oSTeoporosis
Acronym: SAFEST
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC31/23/0370
Record Dates: First submitted 2025-01-06; First posted 2025-01-09 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Postmenopausal Osteoporosis
Keywords: Postmenopausal osteoporosis; strategy; denosumab; zoledronate; rebound; withdrawal
MeSH Terms: conditions — Osteoporosis, Postmenopausal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive biomarkers-guided arm (Experimental): A second infusion when crosslaps levels reach 300 pg/mL, no later than month-12
  Interventions: Drug: a second infusion of ZOL when crosslaps levels reach 300 pg/mL
- Standard treatment arm (Active Comparator): Potentially a rescue second infusion at month-12, in case unfavourable outcome (incident osteoporotic fractures) or high risk of unfavourable outcome
  Interventions: Drug: a rescue second infusion at month-12 (standard traitment)

INTERVENTIONS:
Drug: a second infusion of ZOL when crosslaps levels reach 300 pg/mL — a first infusion of ZOL 5 mg, 6 months after denosumab withdrawal (= study start) and a second infusion when crosslaps levels reach 300 pg/mL, no later than month-12
  Arms: Intensive biomarkers-guided arm
Drug: a rescue second infusion at month-12 (standard traitment) — a first infusion of ZOL 5 mg, 6 months after denosumab withdrawal (= study start), and potentially a rescue second infusion at month-12, in case unfavourable outcome (incident osteoporotic fractures) or high risk of unfavourable outcome
  Arms: Standard treatment arm

SUMMARY:
Denosumab (Dmab) is a treatment for postmenopausal osteoporosis. However, its withdrawal is associated with a rebound phenomenon associated with an unexpected increased risk of vertebral fractures. Defining the optimal strategy for Dmab withdrawal is critically needed. Investigator propose an open-label randomized superiority strategy trial to compare the 1-year lumbar densitometric efficacy of biomarkers-driven zoledronate (ZOL) infusion vs standardized ZOL treatment to mitigate rebound phenomenon.

DETAILED DESCRIPTION:
Denosumab (Dmab) is a potent and validated treatment for postmenopausal osteoporosis. However, its withdrawal, especially after reaching therapeutic target, is associated with a rebound phenomenon characterized by: (i) an increase in bone turnover markers levels usually within first 6 months off-treatment, (ii) a decrease in BMD, and (iii) an unexpected increased risk of (multiple) vertebral fractures. Although current experts' recommendations propose a post-Dmab bisphosphonates therapy (such as ZOL) to mitigate rebound phenomenon, the optimal strategy is still matter of debate. Data suggesting a protective effect with bisphosphonates (1 infusion of ZOL or weekly alendronate) are scarce, with discrepancies, and highlight that a substantial proportion of patients experiences rebound-related bone loss despite bisphosphonate therapy. Crosslaps, a bone turnover maker, are available for daily clinical practice and reflect the antiresorptive activity of anti-resorptive drugs such as bisphosphonates. Investigator hypothesize that monitoring crosslaps levels, can help to identify patients requiring more intensive bisphosphonate (additional ZOL infusion) therapy to control the post-Dmab rebound phenomenon.

Investigator propose to compare 2 strategies for Dmab withdrawal in postmenopausal osteoporosis: a standard treatment control group treated with a single ZOL infusion versus a biomarker-guided ZOL group with an additional ZOL infusion in case of insufficient inhibition of bone resorption according to crosslaps.

ELIGIBILITY:
Inclusion Criteria:

* Women with post-menopausal osteoporosis
* And treated with denosumab for at least 2 years and reaching decision of denosumab withdrawal because of achieved therapeutic target defined as no fracture during treatment; no new risk factors; no BMD decrease > 0.03 g/cm² at the spine or hip;
* And with a history of severe fracture or a femoral or lumbar T-score ≤ -2.5 prior denosumab initiation.

Exclusion Criteria:

* Dmab use for bone disease other than post-menopausal osteoporosis.
* Uncontrolled endocrine diseases. Liver failure.
* Use of medication affecting bone metabolism during the last year, including bisphosphonates, teriparatide, romosozumab, Selective Estrogen Receptor Modulators, breast cancer hormonotherapy, glucocorticoids over 5 mg/day.
* Contra-indication to bisphosphonates according to license recommendation including chronic kidney disease with GFR stage > or = G3b. Prior intolerance to zoledronic acid.
* Subjects unable to give an informed consent or to fill the case report form. Subjects under law protection.
* Foreseeable poor compliance with the strategy, alcoholism, toxicomania.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — postmenopausal osteoporosis
Enrollment: 200 (Estimated)
Dates: Start 2025-10-02 (Actual); Primary Completion 2030-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Maintain lumbar bone mineral density (BMD) after 1 year of ZOL | 1 year after inclusion
  The proportion of patients who failed to maintain lumbar BMD after 1 year of ZOL according to the Least Significant Change (LSC) criterion

SECONDARY OUTCOMES:
Maintain hip bone mineral density (BMD) after 1 year of ZOL | 1 year after inclusion
  The proportion of patients who failed to maintain hip BMD after 1 year of ZOL according to the Least Significant Change (LSC) criterion
the changes in hip and lumbar BMD from baseline | Day 0, 1 year after inclusion, 2 year after inclusion
  the changes in hip and lumbar BMD from baseline to 1 year, and from year 1 to year 2 after ZOL, according to the Least Significant Change (LSC) criterion
the changes from baseline in bone turnover markers | 1 year after inclusion, 2 year after inclusion
  Bone turnover markers is a composite measure derived from crosslaps, bone alkaline phosphatase, osteocalcin, amino-terminal propeptide of type 1 procollagen, TRAP5b, dickkopf 1, sclerostin
morphometric vertebral fractures | 1 year after inclusion, 2 year after inclusion
  the number of morphometric vertebral fractures measured by vertebral fracture assessment (VFA) or X-rays, of clinical vertebral fractures and of clinical peripheral fractures
Patients requiring a second ZOL | 1 year after inclusion, 2 year after inclusion
  the proportion of patients requiring a second ZOL infusion across groups.
Relation between biomarker values and densitometry evolution | 3, 6, 9, 12 months after inclusion
  the relation is defined by biomarker values (cross laps) and densitometry evolution measured bu osteodensitometry
Relation between biomarker values and appearance of new vertebral fracture | 3, 6, 9, 12 months after inclusion
  the relation is defined by biomarker values (cross laps) and appearance of new vertebral fracture measured by VFA or X-rays

CONTACTS AND LOCATIONS:
Locations (17):
- France (17):
  - Amiens Hospital, Amiens
  - Bordeaux Hospital, Bordeaux
  - Cahors Hospital, Cahors
  - Dax Hospital, Dax
  - Le Mans Hospital, Le Mans
  - Lille Hospital, Lille
  - Limoges Hospital, Limoges
  - Marseille Hsopital, Marseille
  - Montpellier Hospital, Montpellier
  - Nice Hospital, Nice
  - Orléans Hospital, Orléans
  - Cochin Hospital, Paris
  - Lariboisiere Hospital, Paris
  - Poitiers Hospital, Poitiers
  - Rennes Hospital, Rennes
  - Saint Etienne Hospital, Saint-Etienne
  - Toulouse Hospital, Toulouse